CLINICAL TRIAL: NCT02378012
Title: Project BUCKiPAD: The Evaluation of an iPAD Distribution Program on Anxiety and Depression in Bone and Marrow Transplant Patients
Brief Title: iPad Use in Reducing Anxiety and Depression in Patients Undergoing Bone Marrow Transplant
Acronym: BUCKiPAD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Competing study
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Samantha Jaglowski, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-12207; NCI-2014-00935 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-02-26; First posted 2015-03-04 (Estimated); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Anxiety; Depression; Malignant Neoplasm
MeSH Terms: conditions — Anxiety Disorders; Depression; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GROUP A (participants provide own computer or tablet device) (Active Comparator): A member of the research personnel helps the participants install Netflix, Spotify, and Skype applications on their computers if they wish to do so. Participants will be given subscriptions to each application and usernames for access on days -5 to 10.
  Interventions: Other: Computer-Assisted Intervention; Other: Questionnaire Administration
- GROUP B (Apple BuckiPad) (Experimental): Participants receive an iPad for days -5 to 10. Participants also receive the BuckiPad manual for instructions on how to use the iPad and Netflix, Skype, and Spotify applications. Participants are also directed to the official Apple's iPad user's manual on their device and have questions answered by research personnel on day -5.
  Interventions: Other: Computer-Assisted Intervention; Other: Questionnaire Administration
- GROUP C (no intervention) (No Intervention): Participants do not receive an iPad for days -5 to 10.

INTERVENTIONS:
Other: Computer-Assisted Intervention — Receive access to Netflix, Spotify, and Skype applications
  Arms: GROUP A (participants provide own computer or tablet device); GROUP B (Apple BuckiPad)
Other: Computer-Assisted Intervention — Receive iPad and instruction manuals.
  Arms: GROUP B (Apple BuckiPad)
Other: Questionnaire Administration — Ancillary studies
  Arms: GROUP A (participants provide own computer or tablet device); GROUP B (Apple BuckiPad)

SUMMARY:
This randomized clinical trial studies iPad use in reducing anxiety and depression in patients undergoing bone marrow transplant. A tablet device like the iPad can provide access to music, television, movies, books, and the Internet. It also contains a video conferencing system that can allow patients to communicate with family members and other members of their social support team. With these capabilities, an iPad distribution program may help lessen patient anxiety and depression during a hospital stay. Monitoring iPad use by patients may help doctors better understand how patients use their computers and tablets while in the hospital so that the software and applications of the iPad can be made more useful.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the effect access to an iPad has on anxiety as measured by the Hospital Anxiety and Depression Scale.

SECONDARY OBJECTIVES:

I. Determine how computers and tablets are used by patients who have access to such devices.

OUTLINE: Participants are assigned to Group A or randomized to 1 of 2 groups (Groups B or C).

GROUP A (participants provide their own computer or tablet device): A member of the research personnel helps the participants install Netflix, Spotify, and Skype applications on their computers if they wish to do so. Participants will be given subscriptions to each application and usernames for access on days -5 to 10.

GROUP B (Apple iPad): Participants receive an iPad for days -5 to 10. Participants also receive the BuckiPad manual for instructions on how to use the iPad and Netflix, Skype, and Spotify applications. Participants are also directed to the official Apple's iPad user's manual on their device and have questions answered by research personnel on day -5.

GROUP C: Participants do not receive an iPad for days -5 to 10.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing treatment in the bone marrow transplant (BMT) unit on the 3rd floor of the James Cancer Hospital and Solove Research Institute
* Patients receiving reduced intensity chemotherapy for an allogeneic stem cell transplant

Exclusion Criteria:

* Patients who lack the visual or motor skills necessary to use a tablet device like the Apple iPad

  * Criteria for visual proficiency will be determined by asking the patient: do you have trouble reading a newspaper even with your glasses or contacts (if you wear them); if "yes", they will be excluded
  * Criteria for motor skill proficiency will be determined by asking the patient: do you have any trouble using a television remote control; if "yes", they will be excluded
* Patients who do not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-03-19 (Actual); Primary Completion 2014-09-06 (Actual); Study Completion 2014-09-06 (Actual)

PRIMARY OUTCOMES:
Change in Hospital Anxiety and Depression Scale (HADS)-Anxiety score | Baseline to day 10
  Will be analyzed using an analysis of covariance (ANCOVA) model containing fixed effects of treatment condition (iPAD vs. no iPAD), baseline HADS-Anxiety score, and a random, normally distributed error term. The data will be log-transformed prior to analysis, so all resulting inferences will be based on the geometric mean instead of the arithmetic mean.

SECONDARY OUTCOMES:
Change in HADS depression score | Baseline to day 10
  Will be analyzed using an ANCOVA model containing fixed effects of treatment condition (iPAD vs. no iPAD), baseline HADS-Depression score, and a random, normally distributed error term. The data will be log-transformed prior to analysis, so all resulting inferences will be based on the geometric mean instead of the arithmetic mean.
Change in Profile of Mood States Short Form (POMS-SF) scores | Baseline to day 10
  Will be analyzed using an ANCOVA model containing fixed effects of treatment condition (iPAD vs. no iPAD), baseline POMS-SF score, and a random, normally distributed error term. The data will be log-transformed prior to analysis, so all resulting inferences will be based on the geometric mean instead of the arithmetic mean.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Jaglowski, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu